CLINICAL TRIAL: NCT03246243
Title: Quantitative Assessment of Sucking for Early Diagnosis of Brain Injury in Infants at High Risk
Status: Terminated | Type: Observational
Why Stopped: Difficulties in recruitment.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Winchester Hospital (Unknown)
Responsible Party: Principal Investigator, Christos Papadelis, PhD, Boston Children's Hospital
Other Study IDs: IRB-P00023193
Record Dates: First submitted 2017-06-21; First posted 2017-08-11 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Hypoglycemia; Neonatal Abstinence Syndrome
Keywords: Hypoxic Ischemic Encephalopathy; Bottle Feeding; Hypoglycemia; Neonatal Abstinence Syndrome; Abnormal Neurodevelopment
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypoglycemia; Neonatal Abstinence Syndrome; Bottle Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Preterm infants: Group A will consist of preterm infants born < 37 weeks gestational age. Non-nutritive and nutritive sucking will be assessed using an FDA-approved device (Nfant Feeding Solution) to measure sucking activity. Additionally, those infants who have MRI of the brain for any reason during the course of their hospital admission will also be included in the study and allocated to the appropriate group accordingly. If a subject undergoes any clinically ordered EEG, EMG, MEG, and MRI throughout the duration of their study participation before the age of three then that data will be collected from their medical record. Additionally, any neurodevelopmental testing data completed up to the age of three will be collected.
  Interventions: Device: nfant feeding solution
- Term infants with HIE or at risk of brain injury: Group B will consist of term infants admitted to the NICU for therapeutic hypothermia who are at risk of HIE; admitted with concern for neonatal stroke; seizures of unknown etiology; and those admitted who are at risk of abnormal neurodevelopment such as those with hypoglycemia or NAS. Non-nutritive and nutritive sucking will be assessed using an FDA-approved device (Nfant Feeding Solution) to measure sucking activity. Additionally, those infants who have MRI of the brain for any reason during the course of their hospital admission will also be included in the study and allocated to the appropriate group accordingly. If a subject undergoes any clinically ordered EEG, EMG, MEG, and MRI throughout the duration of their study participation before the age of three then that data will be collected from their medical record. Additionally, any neurodevelopmental testing data completed up to the age of three will be collected.
  Interventions: Device: nfant feeding solution
- Term infants healthy at birth: Group C will consist of healthy term infants from the community and term infants admitted to who had an initial uncomplicated postnatal course that will serve as the control group. Non-nutritive and nutritive sucking will be assessed using an FDA-approved device (Nfant Feeding Solution) to measure sucking activity. Additionally, those infants who have MRI of the brain for any reason during the course of their hospital admission will also be included in the study and allocated to the appropriate group accordingly. If a subject undergoes any clinically ordered EEG, EMG, MEG, and MRI throughout the duration of their study participation before the age of three then that data will be collected from their medical record. Additionally, any neurodevelopmental testing data completed up to the age of three will be collected.
  Interventions: Device: nfant feeding solution

INTERVENTIONS:
Device: nfant feeding solution — The study will record the sucking activity of the hospitalized infants over time, from their first oral sucking session including non-nutritive and nutritive sucking, until discharge, using an FDA-approved device that equips a typical bottle and nipple commonly used in the NICU with a non-invasive sensor to measure sucking activity. Each infant's nutritive and non-nutritive sucking patterns will be measured, and will comprise the 'sucking session' conducted with the bottle sensor.

SUMMARY:
The main goal of this study is to quantitatively assess the sucking and feeding activity of infants at high risk of neurological impairment (preterm infants and term infants at risk of abnormal neurodevelopment) during oral sucking and feeding and correlate it with their underlying neurological impairment for the early diagnosis of brain injury.

DETAILED DESCRIPTION:
This research will address the current lack of objective tools for the reliable assessment of oral sucking and feeding in clinical practice, and the insufficient evidence that relates early measures of abnormal sucking activity with the underlying neurological impairment.

The main goal of this study is to quantitatively assess the sucking and feeding activity of infants at high risk of neurological impairment (preterm infants and term infants at risk of abnormal neurodevelopment) during oral sucking and feeding and correlate it with their underlying neurological impairment for the early diagnosis of brain injury. We aim to study three groups of infants who are inpatients on the Neonatal Intensive Care Unit (NICU) at Boston Children's Hospital (BCH), the NICU or Newborn Nursery at Beth Israel Deaconess Medical Center (BIDMC), the Special Care Nursery (SCN) or Newborn Nursery at Winchester Hospital as follows: (i) group A consisting of preterm infants (gestational age of <37 weeks), (ii) group B consisting of term infants admitted to the NICU at BCH and BIDMC for therapeutic hypothermia who are at risk of developing hypoxic ischemic injury (HIE); admitted with concern for neonatal stroke; seizures of unknown etiology; and those admitted to the NICU, SCN or Newborn Nursery at BCH, BIDMC and Winchester Hospital at risk of abnormal neurodevelopment such as those with hypoglycemia or neonatal abstinence syndrome (NAS) and; (iii) group C consisting of healthy term infants admitted to the NICU, SCN or nursery who had an initial uncomplicated postnatal course that will serve as the control group. Additionally, those infants who have MRI of the brain for any reason during the course of their hospital admission will also be included in the study and allocated to the appropriate group accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with GA<37 weeks
* Term infants with GA>37 weeks and at risk of brain injury
* Healthy term infants with GA= 37-41 weeks, appropriate birth weight, 5 minute Apgar score>7, and an initial uncomplicated postnatal course

Exclusion Criteria:

* major congenital anomalies
* craniofacial malformation
* short bowel syndrome

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants at risk of brain injury; Term infants at risk of brain injury; and Healthy term infants.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Difference in sucking activity of infants with brain injury | Approximately one year through study completion
  Primary outcome will be an assessment of the sucking activity of infants with brain injury and infants without brain injury, using an FDA-approved device for sucking assessment.

SECONDARY OUTCOMES:
Sucking activity of infants and brain connectivity | Approximately three years through study completion
  The functional and structural connectivity of the brain areas involved in sucking and feeding in infants with brain injury will be assessed reviewing the results of clinically ordered neuroimaging and neurodevelopmental tests.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Papadelis, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No